CLINICAL TRIAL: NCT01087593
Title: Hormonal Replacement Therapy Does Not Affect Self-estimated Pain or Experimental Pain Responses in Postmenopausal Women Suffering From Fibromyalgia: A Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Estrogens Effect on Pain in Postmenopausal Women Suffering of Fibromyalgia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to ethical concerns regard to the results from the WHI study
Sponsor: Ostergotland County Council, Sweden (Other)
Responsible Party: Mats Hammar, Ostergotland County Council
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 151 662/01
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2001-09

CONDITIONS: Fibromyalgia
Keywords: estrogen; substitution; pain; hormonal levels; quantitative sensory testing
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Estradiol; Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with transdermal 17β-estradiol (Experimental)
  Interventions: Drug: 17β-estradiol
- Control (Placebo Comparator)
  Interventions: Drug: 17β-estradiol

INTERVENTIONS:
Drug: 17β-estradiol — Transdermal administration(50 ug daily)for a period of ten weeks with additional treatment of medroxyprogesterone (10mg daily) for the last two weeks
  Other Names: Evorel; provera

SUMMARY:
In order to evaluate the potential effects of estrogen treatment in postmenopausal women with fibromyalgia, the investigators used quantitative sensory tests before and after eight weeks of estrogen treatment as compared with placebo treatment.

DETAILED DESCRIPTION:
Fibromyalgia is a condition that preferentially affects women. Sex hormones, and in particular estrogens, have been shown to affect pain processing and pain sensitivity, and estrogen deficit has been considered a potential promoting factor for fibromyalgia. However, the effects of estrogen treatment in patients suffering from fibromyalgia have not been studied. Twenty-nine postmenopausal women were randomized to either eight weeks of treatment with transdermal 17β-estradiol (50 ug daily) or placebo according to a double-blind protocol. A self-estimation of pain, a set of quantitative sensory tests measuring thresholds to temperature, thermal pain, cold pain and pressure pain, and a cold pressor test were performed at three occasions: before treatment, after eight weeks of treatment, and twenty weeks after cessation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between 49-60 years
* Body mass index (BMI) of < 30
* Met the ACR-90 criteria for the diagnosis of fibromyalgia
* Postmenopausal state since at least six months
* Not been using any hormonal treatments for the past three months
* Had normal mammography screenings

Exclusion Criteria:

* Using psychotropic drugs or having a history of thromboembolism
* Diabetes mellitus, polyneuropathy, chronic liver disease,
* Alcohol or substance abuse, hemoglobinopathy,
* Endometrial adenomatous hyperplasia, or malignancy.
* Presence of untreated hypertension (>160/95).
* Undiagnosed vaginal bleedings

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2001-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Pain thresholds and pain tolerance | Before and after eight weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mats Hammar, MD, prof, Principal Investigator — University Hospital, Linkoeping
Locations (1):
- University hospital in Linköping, Linköping, Sweden

REFERENCES:
- [Derived] Stening KD, Eriksson O, Henriksson KG, Brynhildsen J, Lindh-Astrand L, Berg G, Hammar M, Amandusson A, Blomqvist A. Hormonal replacement therapy does not affect self-estimated pain or experimental pain responses in post-menopausal women suffering from fibromyalgia: a double-blind, randomized, placebo-controlled trial. Rheumatology (Oxford). 2011 Mar;50(3):544-51. doi: 10.1093/rheumatology/keq348. Epub 2010 Nov 14. PMID 21078629